CLINICAL TRIAL: NCT04860037
Title: Micromegaly and Discrepancy Between Growth Hormone and IGF1 at the Diagnosis and Follow-up of Acromegalic Patients : What About Their Consequences ?
Brief Title: Micromegaly and Discrepancy Between Growth Hormone and IGF1 at the Diagnosis and Follow-up of Acromegalic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0229
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Acromegaly
Keywords: Endocrinology; Acromegaly; Discrepancy; Complications
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The diagnosis and the follow-up of acromegalic patients are based on the mesurement of Growth hormone (GH) and IGF1 rates. However, the literature described some cases of patient for whom the investigators observed a discrepancy between GH and IGF1 rates. Since the acromegaly is a rare disease and this phenomenon concerns about 30% of these patients, there is a lack of investigations about consequences that this discordance may induces. In this study, the investigators aimed at assessing if patients with discordance between GH and IGF1 rates present a different risk of recurrence and complications related to acromegaly, from patients with concordant results.

ELIGIBILITY:
Inclusion criteria:

* Acromegaly followed up in one of the center (Montpellier, Nimes or Béziers hospital, independent endocrinologist) between 2010 and 2021
* Age over 18 years old
* Measurement of GH and IGF1 rates at the last visit control available

Exclusion criteria:

* Lost to follow-up
* Status about complications related to acromegaly unknown

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult acromegalic patient followed up in the Occitanie region (independent endocrinologist ou working in hospital of Montpellier, Nimes or Béziers)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of complications and/or recidivism related to acromegaly | day 1
  The investigators check in the patient file if there is complications or pathology recidivism detected at the last full check-up of the disease, assessed by blood-control and complementary exams

SECONDARY OUTCOMES:
Disease's specificity | day 1
  The investigators collected datas about disease's diagnosis (IRM characteristic, GH/IGF1 rates, clinical presentation) to evaluate if there is a different initial presentation between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle RAINGEARD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC